CLINICAL TRIAL: NCT06474468
Title: A Phase IB /II, Multicenter, Open-Label Study of Safety, Tolerability and Efficacy of SHR-A2102 for Injection With Adebrelimab With or Without Other Antitumor Therapy in Advanced or Metastatic Esophageal Cancer
Brief Title: A Trial of SHR-A2102 With Adebrelimab With or Without Other Antitumor Therapy in Advanced or Metastatic Esophageal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-203
Record Dates: First submitted 2024-06-06; First posted 2024-06-25 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-06

CONDITIONS: Advanced or Metastatic Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group A/B (Experimental): A：SHR-A2102+Adebrelimab B：SHR-A2102+Adebrelimab+Cisplatin
  Interventions: Drug: SHR-A2102；Adebrelimab；Cisplatin

INTERVENTIONS:
Drug: SHR-A2102；Adebrelimab；Cisplatin — Drug: SHR-A2102 Administration by intravenous infusion for a cycle of 3 weeks.
  Drug: Adebrelimab Administration by intravenous infusion for a cycle of 3 weeks.
  Drug: Cisplatin Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and efficacy of SHR-A2102 with Adebrelimab with or without other Antitumor Therapy in Advanced or Metastatic Esophageal Cancer. To explore the reasonable dosage of SHR-A2102 for Advanced or Metastatic Esophageal Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to give informed consent, have signed informed and able to comply with the treatment plan to visit the tests and other procedural requirements；
2. The age of signing the informed consent is 18 -70 years, regardless of gender；
3. Provide archived or fresh tumor tissue for vendor test;
4. At least one measurable lesion according to RECIST v1.1 criteria；
5. Subjects with pathology confirmed locally advanced unresectable or metastatic esophageal squamous cell carcinoma;
6. The ECOG score is 0 or 1；
7. Expected survival ≥12 weeks
8. Good level of organ function
9. Male subjects whose partners are women of childbearing age and female subjects who are fertile are required to use highly effective contraceptive methods.

Exclusion Criteria:

1. Inadequately treated central nervous system metastases or the presence of uncontrolled or symptomatic active central nervous system metastases；
2. Patients with uncontrolled tumor-related pain as determined by the investigator.
3. Moderate or severe ascites with clinical symptoms (i.e., those who required therapeutic puncture or drainage within 2 weeks before the study treatment, and only those who showed a small amount of ascites without clinical symptoms could be included in the study); Unable to control or moderate or higher amounts of pleural effusion or pericardial effusion
4. A history of gastrointestinal perforation and/or fistula within 6 months prior to initial medication, or significant tumor invasion of adjacent organs (large arteries or trachea, etc.), resulting in a higher risk of bleeding or fistula
5. Have antitumor therapy was received 4 weeks before the start of the study；
6. Have previously received antiboy-coupled drugs containing topoisomerase I inhibitors
7. Systemic antitumor therapy was received 4 weeks before the start of the study
8. Treatment with CYP3A4, CYP2D6, P-gp, or BCRP booster or inducer is less than 5 drug half-lives from the date of first administration
9. Surgical procedures requiring tracheal intubation and general anesthesia were performed within 28 days prior to the initial study, diagnostic or superficial surgery was performed within 7 days prior to the initial study, or elective surgery was expected during the trial period;
10. Perform non-chest radiation therapy with >30Gy within 28 days before dosing, chest radiation therapy with >30Gy within 24 weeks before first dosing, and radiation therapy with ≤30Gy within 14 days before first dosing
11. Toxicity and/or complications of previous antitumor therapy did not return to NCI-CTCAE level ≤1 or exclusion criteria
12. Live attenuated vaccines were used within 28 days prior to initial study administration or during the expected study treatment；
13. Systemic immunosuppressive therapy was administered within 14 days prior to the first study
14. Subjects with known or suspected interstitial pneumonia;
15. In the first study, a single blood loss ≥50ml or a cumulative daily blood loss ≥300m occurred within 1 month before medication
16. Subjects with severe cardiovascular and cerebrovascular disease;
17. Arterial/venous thrombosis events, such as deep vein thrombosis and pulmonary embolism, occurred within 3 months prior to initial administration
18. Had been diagnosed with any other malignancy
19. Subjects who had a severe infection within 28 days prior to the first dose
20. Active hepatitis B or active hepatitis C
21. Patients with active pulmonary tuberculosis within 1 year prior to enrolment
22. History of immune deficiency
23. Severe allergic reactions are known to occur in individuals allergic to any component of SHR-A2102, SHR-1316, or other monoclonal antibody/fusion protein drugs
24. Per the investigator's judgment, there are any other circumstances that may increase the risk of participating in the study, interfere with the study results, or make participation in the study inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
RP2D | through phase IB completion, an average of 1 years
  RP2D will be determined on the basis of evaluation on safety, PK, efficacy data in Phase IB stages；
Incidence and severity of AE(DLT)： | from Day1 to 90 days after last dose
  According to NCI-CTCAE v5.0 evaluation criteria from Day 1 to 90 days after last dose；
ORR： | 18 months after the last subject was enrolled in the group
  efficacy was assessed every 6 weeks within 48 weeks and every 9 weeks after 48 weeks s as determined by RECIST1.1

SECONDARY OUTCOMES:
DCR | 18 months after the last subject was enrolled in the group
  Since C1D1 every 6 weeks within 48 weeks and every 9 weeks after 48 weeks, and the proportion of subjects whose best response was PR or CR or SD as determined by RECIST1.1；
DOR | 18 months after the last subject was enrolled in the group
  Since C1D1 every 6 weeks within 48 weeks and every 9 weeks after 48 weeks, and the proportion of subjects whose best response was PR or CR or SD as determined by RECIST1.1；
PFS(Investigator evaluation) | 18 months after the last subject was enrolled in the group
  Since C1D1 every 6 weeks within 48 weeks and every 9 weeks after 48 weeks, and the proportion of subjects whose best response was PR or CR or SD as determined by RECIST1.1；
OS(Investigator evaluation) | 18 months after the last subject was enrolled in the group
  Since C1D1 and death from any cause；

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided